CLINICAL TRIAL: NCT01900067
Title: An Open-Label, Multicenter, Randomised, Controlled Study to Evaluate the Efficacy and Safety of the BARRIER® EasyWarm Active Self-Warming Blanket Used for Continuous Active Warming to Prevent General Anaesthesia Induced Hypothermia During the Perioperative Surgical Period
Brief Title: Study to Evaluate Safety and Efficacy of Blanket Used to Prevent Anesthesia Induced Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MD12-001
Record Dates: First submitted 2013-07-08; First posted 2013-07-16 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2014-12

CONDITIONS: Anesthesia Induced Hypothermia; Inadvertent Perioperative Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active warming (Active Comparator): BARRIER® EasyWarm Active Self-Warming Blanket
  Interventions: Device: BARRIER® EasyWarm Active Self-Warming Blanket
- Control (No Intervention): no active warming, standard of care

INTERVENTIONS:
Device: BARRIER® EasyWarm Active Self-Warming Blanket
  Other Names: active warming
  Arms: Active warming

SUMMARY:
The investigation was designed as an Open-Label, Multicenter, Randomised, Controlled Investigation to Evaluate the Efficacy and Safety of the BARRIER® EasyWarm Active Self-Warming Blanket Used for Continuous Active Warming to Prevent General Anaesthesia Induced Hypothermia During the Perioperative Surgical Period. Null hypothesis (H0): There is no difference between the two study populations (interventional treatment group versus control treatment group) regarding the average of core body temperature measurements during the perioperative phase.Alternative hypothesis (H1): The average of core body temperature measurements during the perioperative phase is significantly higher in the interventional group compared to that of the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Both men and women are included into the study
2. Subjects' age: Subjects must be at least 18 years old to be included into the study
3. Type of anaesthesia: Only subjects receiving general anaesthesia are included into the study
4. Type of surgery: Subjects undergoing only the following three types of surgical procedures (i.e. inclusive of laparoscopic procedures) are included into the study:

   * Gynaecological
   * Orthopaedic
   * Ear, nose and throat (ENT)
5. Length of surgery: Subjects scheduled for a surgery with a minimum length of 30 minutes and maximum length of 120 minutes
6. Temperature: Subjects should have a tympanic temperature measurement equal to or greater than 36.0 degrees Celsius when first measured in the preoperative setting the same day as the surgical procedure and before randomisation
7. Informed Consent Form (ICF): The subject must be able to understand and sign an ICF
8. Method of temperature assessment: The subject must be able to receive temperature assessments via a tympanic thermometer
9. Preoperative warming: Subject's scheduled surgical procedure must allow time to be warmed with a fully activated study Investigational Device (ID), at least 30 minutes prior to induction of general anaesthesia
10. Follow up: The subject must be able to complete a health outcomes questionnaire for follow up 24 hours (+/- 6 hours) after removal of the ID

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) Physical Status Classification rating: Subjects with a ASA rating of 4 or greater are excluded from the study
2. Comorbidity: Known Diabetes with an HbA1c of more than 6 %
3. Temperature: Subjects with a tympanic temperature measurement below 36.0 degrees Celsius taken in the preoperative setting
4. Medical history: Subject reports relevant medical history (e.g., neuropathy, peripheral vascular disease, or other) that presents risk to/of:

   1. The subject's normal temperature regulation or
   2. Perception of external temperature or
   3. Subcutaneous lipoatrophy
5. Medication: Current use of concomitant medications that present relevant risk to/of:

   1. The subject's normal temperature regulation or
   2. Perception of external temperature or Clinical Investigation Plan with Integrated Amendments 01 and 02, MD12-001, final, 14-Jan-2013 5(32)
   3. Subcutaneous lipoatrophy or
   4. All locoregional and neuroaxial blocks
6. Other:

   1. Presence of skin and soft tissue disorders in areas covered directly by the ID (e.g., pressure ulcers, clinically significant psoriasis, dermatitis or any other interruption of skin integrity that would be affected by direct heat)
   2. Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Torossian, Prof, Principal Investigator — Universitätsklinikum Gießen und Marburg; Johan Raeder, Prof, Principal Investigator — OUS-Ullevål; Karin Geertsen, Dr, Principal Investigator — Hallands sjukhus Varberg; Bengt Horn af Åminne, Dr, Principal Investigator — Aleris Specialistvård, Motala; Elke Van Gerven, Dr, Principal Investigator — UZ Leuven Gasthuisberg; Marc Van de Velde, Prof., Study Chair — UZ Leuven Gasthuisberg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Warming | Control
Started | 134 | 137
Completed | 122 | 124
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Warming | Control | Total
Number analyzed (Participants) | 122 | 124 | 246
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 46.5 (15.3) | 45.6 (14.8) | 46.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 96 | 188
  Male | 30 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: The Difference in the Arithmetic Mean of Core Body Temperature Measurements During the Perioperative Phase Between the Interventional Treatment Group and the Control Treatment Group
Description: The subject's core body temperature at any time point is approximated by the arithmetic mean of three repeated tympanic temperature measurements every 15 minutes during the perioperative period
Time Frame: temperature measurments during pre,-intra and postoperative period, on average 1-5 hours, depending on the surgical intervention.
Measure: Mean (95% Confidence Interval); unit: Degree Celsius (°C)
Arm/Group | Active Warming | Control
Number analyzed (Participants) | 122 | 124
Degree Celsius (°C) | 36.52 [36.15 to 36.89] | 36.34 [36.0 to 36.74]

ADVERSE EVENTS:
Arm/Group | Active Warming | Control
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/137
Other Adverse Events (participants affected / at risk) | 23/134 | 0/137
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Warming (N=134) | Control (N=137)
Redness of skin (Skin and subcutaneous tissue disorders) | 23 (23) | 0 (0) — All adverse device effects were of the type redness of skin under one or more of the warmers of the device. Once the device was removed the redness vanished quickly without further treatment. Redness was judged to be caused by local vasodilatation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement state that sponsor is the owner of all results. The Investigator may perform a secondary publication from an individual investigation site without disclosing confidential information received from sponsor after the multi-center publication or within 12 months after termination of the investigation if no such multi-centre publication takes place.